CLINICAL TRIAL: NCT00331799
Title: A Pilot Study of Duloxetine in Psychological Resilience and Its Correlation With Blockade of Serotonin and Norepinephrine Transporter
Brief Title: Pilot Study of Duloxetine in Psychological Resilience
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008715
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Results first posted 2013-08-02 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-06

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Pharmacotherapy; Duloxetine
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): Open label treatment with Duloxetine for 8 weeks with dosing from 30-60 mg.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — Open label treatment with Duloxetine for 8 wks. Dose 30-60 mg.
  Other Names: Cymbalta

SUMMARY:
The purpose of this study is to explore benefits of duloxetine in enhancing psychological resilience and to understand the relevance of inhibiting of both serotonin (5HT) and norepinephrine (NE)to therapeutic responses.

DETAILED DESCRIPTION:
This is an investigator-initiated, single-site study consisting of 8 weeks of open-label, fixed-dose treatment with duloxetine (30mg-60mg/day) in patients with Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* ages 18-65
* primary diagnosis of MDD based on Diagnostic Standard Manual(DSM-IV) criteria and assessed by the MINI International Neuropsychiatric Interview
* Montgomery-Asberg Depression Rating Scale (MADRS)score of at least 20 on baseline
* Minimum Clinical Global Impressions of Severity (CGS) severity score of 4
* Ability to provide written consent form
* A negative serum pregnancy test for women of childbearing potential

Exclusion Criteria:

* Current DSM-IV diagnosis of bipolar disorder, schizophrenia or other psychotic disorder, mental retardation or other pervasive developmental disorder or cognitive disorder due to a general medical condition
* History of substance abuse or dependence within the last 6 months
* Suicide risk or serious suicide attempt within the last year
* Clinically significant medical condition or laboratory abnormality
* Women of childbearing potential who are unwilling to practice an acceptable method of contraception
* Subjects needing concurrent use of psychotropic medications
* History of sensitivity to duloxetine
* History of failure to respond to an adequate trial of duloxetine (at least 60mg/day for 4 weeks)
* Subjects taking monoamine oxidase inhibitors (MAOIs)
* Subjects with uncontrolled narrow-angle glaucoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Bymaster FP, Dreshfield-Ahmad LJ, Threlkeld PG, Shaw JL, Thompson L, Nelson DL, Hemrick-Luecke SK, Wong DT. Comparative affinity of duloxetine and venlafaxine for serotonin and norepinephrine transporters in vitro and in vivo, human serotonin receptor subtypes, and other neuronal receptors. Neuropsychopharmacology. 2001 Dec;25(6):871-80. doi: 10.1016/S0893-133X(01)00298-6. PMID 11750180
- [Background] Charney DS. Psychobiological mechanisms of resilience and vulnerability: implications for successful adaptation to extreme stress. Am J Psychiatry. 2004 Feb;161(2):195-216. doi: 10.1176/appi.ajp.161.2.195. PMID 14754765
- [Background] Connor KM, Davidson JR. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. 2003;18(2):76-82. doi: 10.1002/da.10113. PMID 12964174
- [Background] Davidson J, Watkins L, Owens M, Krulewicz S, Connor K, Carpenter D, Krishnan R, Nemeroff C. Effects of paroxetine and venlafaxine XR on heart rate variability in depression. J Clin Psychopharmacol. 2005 Oct;25(5):480-4. doi: 10.1097/01.jcp.0000177547.28961.03. PMID 16160626
- [Background] Gilmor ML, Owens MJ, Nemeroff CB. Inhibition of norepinephrine uptake in patients with major depression treated with paroxetine. Am J Psychiatry. 2002 Oct;159(10):1702-10. doi: 10.1176/appi.ajp.159.10.1702. PMID 12359676
- [Background] Nemeroff CB, Schatzberg AF, Goldstein DJ, Detke MJ, Mallinckrodt C, Lu Y, Tran PV. Duloxetine for the treatment of major depressive disorder. Psychopharmacol Bull. 2002 Autumn;36(4):106-32. PMID 12858150

RESULTS

PARTICIPANT FLOW:
Groups:
- Open Label Treatment With Duloxetine: Open label treatment with Duloxetine for 8 weeks with dosing from 30-60 mg / day .
Period: Overall Study
Arm/Group | Open Label Treatment With Duloxetine
Started | 18
Completed | 15
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Sedation | 1

BASELINE CHARACTERISTICS:
Groups:
- Open Label Treatment: Open label treatment with Duloxetine for 8 weeks with dosing from 30-60 mg.
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 43.44 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Connor Davidson Resilience Scale (CD-RISC) From Baseline to 8 Weeks
Description: CD-RISC has been psychometrically validated, studied in the general population, as well as in clinical samples. Changes in CD-RISC score have been found to be sensitive to the effect of treatment, and impaired resilience has been demonstrated in subjects with depression relative to normal controls using this scale (Connor and Davidson, 2003). The total score ranges from 0-100, with higher scores indicating greater resilience.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Duloxetine: Open label treatment with Duloxetine for 8 weeks with dosing from 30-60 mg.
Arm/Group | Duloxetine
Number analyzed (Participants) | 18
units on a scale | 52.62 (16.61)
Statistical Analysis 1: Comparison: Duloxetine; Wilcoxon Signed Rank test on the difference between the baseline and endpoint score on the CD-RISC; Test type: Superiority or Other; p = 0.00365, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Open Label Treatment
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No